CLINICAL TRIAL: NCT04961762
Title: Effect of a Navigator Program on Post-Hospital Outcomes for Homeless Adults: A Pragmatic Randomized Controlled Trial
Brief Title: Navigator Program for Homeless Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21-058
Record Dates: First submitted 2021-06-20; First posted 2021-07-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-04

CONDITIONS: Homeless Persons; Case Management; Primary Care; Hospital Readmission

STUDY DESIGN:
Intervention Model Description: Intervention: specialized homeless-specific case management services starting during hospitalization and continuing for approximately 3 months after discharge. Usual care: treatment as usual, without access to specialized homeless-specific case management services.
Who Masked: Outcomes Assessor
Masking Description: Research staff who conduct 30-day follow-up interview with participant are masked to participant's assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigator Program (Experimental): In addition to receiving Standard Care, participants in the intervention arm will be assigned to a Homeless Outreach Counsellor. The Homeless Outreach Counsellor will connect with the participant as soon as possible during the admission and will provide support during the hospital admission and for approximately 90 days after hospital discharge.
  Interventions: Other: Navigator Program
- Standard Care (No Intervention): Standard Care consists of support from Care Transition Facilitators who work with patients during their hospital stay to arrange discharge plans and make follow-up arrangements. Care Transition Facilitators do not routinely work with patients after hospital discharge. As part of the routine discharge process, the health care team provides patients with medical recommendations, appointments for follow-up care as needed, a written discharge summary, and prescriptions as needed. If the patient has an identified primary care provider, a copy of the discharge summary is sent electronically to the primary care provider.

INTERVENTIONS:
Other: Navigator Program — The main role of the Homeless Outreach Counsellor is to support continuity and comprehensiveness of care by helping participants follow their post-discharge plans and facilitating strong links with community-based health and social services. The Homeless Outreach Counsellor also helps address specific needs of participants, develop comprehensive care plans with members of patient's multidisciplinary circle of care, and facilitate the transition of clients to long-term community-based health and social services.
  Arms: Navigator Program

SUMMARY:
Individuals experiencing homelessness often have complex health and social needs. This population also faces disproportionate systemic barriers to accessing health care services and social supports, such as not having primary care providers, needing to meet other competing priorities, and difficulties affording medications. These barriers contribute to discontinuities in care, poor health outcomes, and high acute healthcare utilization after hospitalization among this population. This randomized controlled trial aims to evaluate the effect of a case management intervention (the Navigator program) for individuals experiencing homelessness who have been admitted to hospital for medical conditions. This study will examine outcomes over a 180-day period after hospital discharge, including follow-up with primary care providers, acute healthcare utilization, quality of care transitions, and overall health.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have an unplanned admission for any medical cause to the General Internal Medicine service, any Medicine subspecialty service, the Cardiac Intensive Care Unit, and the Medical Surgical Intensive Care Unit
* Identified as being homeless at the time of admission or anytime during the index hospital admission. This includes patients who are: unsheltered (absolutely homeless and living on the streets or in places not intended for human habitation), emergency sheltered (staying in overnight shelters for people who are homeless, as well as shelters for those impacted by family violence), or provisionally accommodated (whose accommodation is temporary or lacks security of tenure).

Exclusion Criteria:

* Unable to provide informed consent to the study
* Previously received services from the Homeless Outreach Counsellor within 90 days of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Follow-Up with Primary Care Provider (PCP) | Within 14 Days of Discharge
  Occurrence of a follow-up visit with a PCP (family physician or nurse practitioner). In-person encounters (e.g., ambulatory clinics, shelter clinics, and community health centers), virtual encounters (with video), and phone calls (without video) will be considered as follow-up visits. These modes of PCP follow-up are consistent with those outlined by quality standards from Health Quality Ontario. The investigators will ascertain PCP follow-up through: 1) participant self-report at the 30-day interview, 2) PCP office confirmation, and 3) administrative databases (OHIP and Community Health Center Databases at ICES).
  PCP follow-up documented in any of the three data sources will be considered sufficient to meet the primary outcome criterion.

SECONDARY OUTCOMES:
Composite All-Cause Hospital Readmission or Mortality | Within 30, 90, and 180 Days of Discharge
  Hospital readmissions will be ascertained from the 30-day interview and administrative databases at ICES. Mortality data will be collected from hospital charts, follow-up with community contacts, or administrative databases at ICES. (Hospital readmissions exclude elective or scheduled admissions, labor and delivery visits, and transfers between services [i.e., from medicine to psychiatry] within the hospital.)
Number of Emergency Department Visits | Within 30, 90, and 180 Days of Discharge
  Number of emergency department visits will be ascertained from the 30-day interview and administrative databases at ICES.

OTHER OUTCOMES:
Leave Against Medical Advice | During Index Admission
  Ascertained from discharge chart review
Connection to Case Manager | At 30-Day Follow-Up Interview
  Connection to a case manager after hospital discharge will be assessed only among participants who report no contact with a case manager in the 30 days prior to their baseline interview.
Attendance of non-PCP Health Care Appointment | Within 180 Days of Discharge
  Non-PCP health care appointments are defined as appointments with any medical specialist or health care provider other than the participant's family physician or nurse practitioner. Only appointments documented in the discharge summary will be assessed for attendance. Attendance will be ascertained by contacting the health care provider.
Self-Reported Experience of Care Transition | At 30-Day Follow-Up Interview
  Ascertained with the Care Transitions Measure-3 (CTM-3). The CTM-3 is an abbreviated version of the original CTM-15, which measures the extent to which the healthcare team accomplished essential care processes in preparing the patient for discharge and participating in post-hospital self-care activities.
  The CTM-3 consists of 3 items with a 4-point scale with responses ranging from "Strongly Disagree" (1) to "Strongly Agree" (4) to the following questions:
  * During this hospital stay, staff took my preferences into account in deciding what my healthcare needs would be when I left.
  * When I left the hospital, I had a good understanding of the things I was responsible for in managing my health.
  * When I left the hospital, I clearly understood the purpose for taking each of my medications
  Items are scored by summing the responses and then linear transforming to a 0-100 range. Higher scores indicate better self-reported experience of care transition.
Number of Days in Hospital | Within 30, 90, and 180 Days of Discharge
  Number of days in hospital will be ascertained from the 30-day interview and administrative databases at ICES. (Days in hospital exclude elective or scheduled admissions and labor and delivery visits.)
Change in Health Status | Baseline and At 30-Day Follow-Up Interview
  Ascertained with the EQ-5D-3L (EuroQol-5 Dimensions-3 Levels). The EQ-5D-3L is a generic measure of health-related quality of life that has been widely used among the homeless population. The EQ-5D-3L includes five 3-level items concerning mobility, self-care, usual activities, pain/discomfort, and anxiety/depression that are weighted to produce a single utility score between 0 and 1. The Visual Analog Scale (VAS) of the EQ-5D-3L will also be included, which will allow participants to rate their overall health, mental health, and physical health from 0 to 100.
Change in Competing Priorities | Baseline and At 30-Day Follow-Up Interview
  Ascertained with the RAND Course of Homelessness Scale. Developed specifically for the homeless population, the RAND scale is a 5-item index of self-reported difficulty in meeting the following subsistence needs over the past 30 days: frequency of difficulty in finding shelter, enough to eat, clothing, a place to wash, and a place to use the bathroom. Possible responses to each item are never (1), rarely (2), sometimes (3), or usually (4) with total scores between 5-20. Higher scores indicate more difficulty in meeting subsistence needs.
Time to Composite All-Cause Hospital Readmission or Mortality | Within 180 Days of Discharge
  Time to all-cause hospital readmission or mortality is defined as the number of days from hospital discharge to the first all-cause hospital readmission or mortality during the 180-day observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen W Hwang, MD, MPH, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Participants will not have consented to allow for IPD to be shared with other researchers outside of the present day.

REFERENCES:
- [Derived] Liu M, Pridham KF, Jenkinson J, Nisenbaum R, Richard L, Pedersen C, Brown R, Virani S, Ellerington F, Ranieri A, Dada O, To M, Fabreau G, McBrien K, Stergiopoulos V, Palepu A, Hwang S. Navigator programme for hospitalised adults experiencing homelessness: protocol for a pragmatic randomised controlled trial. BMJ Open. 2022 Dec 14;12(12):e065688. doi: 10.1136/bmjopen-2022-065688. PMID 36517099

DOCUMENTS (2):
  • Study Protocol (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT04961762/Prot_003.pdf
  • Statistical Analysis Plan (2025-07-29): https://cdn.clinicaltrials.gov/large-docs/62/NCT04961762/SAP_005.pdf